CLINICAL TRIAL: NCT00569426
Title: An Open-label, Randomised, Multi-centre Cross-over Trial in Diabetes Patients Evaluating Preference, Injection Pressure, Pain Perception and Handling When Injections Are Performed With Two Different Needles i.e. NovoFine® 32 Gauge Tip x 6mm and NovoFine® 30 Gauge x 8mm Using a FlexPen® Disposable Insulin Injection Pen
Brief Title: Evaluating the Use of Two Different Needles in Subjects With Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEEDLEN-1637
Record Dates: First submitted 2007-12-04; First posted 2007-12-07 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NovoFine® needle 6 mm
Device: NovoFine® needle 8 mm

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare two needle types when used with a disposable insulin injection pen in the everyday life setting of an insulin treated patient with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities
* Diagnosed type 1 or type 2 diabetes
* Treated with insulin

Exclusion Criteria:

* Previous participation in this trial
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* Any disease or condition which the investigator feels would interfere with the trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2005-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Overall needle preference | after 2-3 weeks of treatment

SECONDARY OUTCOMES:
Injection pressure
Pain perception
Handling and acceptance of needles

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (10):
- United Kingdom (10):
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, Church Village
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Haywards Heath
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, Penarth
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Sheffield

REFERENCES:
- [Result] McKay M, Compion G, Lytzen L. Pain Perception, Patient Preference, Injection Pressure and Handling with NovoFine® 32G x 6mm Versus 30G x 8mm Needle. ADA 2006; : 1968-PO
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com